CLINICAL TRIAL: NCT06436859
Title: Phd Student Msc Midwifery Öznur HAYAT ÖKTEM
Brief Title: The Effect of Stress Ball on Labor Pain, Anxiety and Satisfaction in Labor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Öznur Hayat Öktem (Other)
Responsible Party: Sponsor-Investigator, Öznur Hayat Öktem, PhD student, Gulhane School of Medicine
Organization: Gulhane School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Hayatoktem03
Record Dates: First submitted 2024-05-15; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Pregnancy; Labor
Keywords: Stress ball; labor pain; anxiety; satisfaction
MeSH Terms: conditions — Labor Pain; Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): Stress ball group
  Interventions: Behavioral: stress ball group
- Control group (No Intervention): Routine care

INTERVENTIONS:
Behavioral: stress ball group — According to randomization, pregnant women in the intervention group will receive "stress ball therapy" during labor.
  Arms: Experiment

SUMMARY:
The aim of this study was to determine the effect of stress ball use during labor on labor pain, anxiety and satisfaction levels in women admitted to Karabük Training and Research Hospital for delivery.

H1 Using the Stress Ball in Labor reduces labor pain. H2 Using the Stress Ball in Labor Reduces Anxiety H3 Use of Stress Ball in Labor increases labor satisfaction.

DETAILED DESCRIPTION:
Birth is accepted as one of the physiological behaviors that have existed since the beginning of mankind and whose formation cycle has not changed. Birth is a health condition that many women desire at some point in their lives. While birth is a normal physiological process and should be an important tool for happiness, it also carries risks such as pain, suffering and discomfort. For this reason, one of the first thoughts a pregnant woman has about childbirth is labor pain. Birth pain is a central and universal part of a woman birth experience.Causes of labor pain include psychological factors such as fear and anxiety, previous experiences, birth environment, lack of information and inadequate support, as well as physical causes such as uterine contractions, cervical dilatation and effacement. Anxiety and tension experienced by pregnant women during the labor process can slow down the progress of labor. Anxiety also reduces women self-confidence, and pregnant women perceive themselves as inadequate and incompetent. Anxiety experienced during labor leads women to cesarean section at their own request.

Utilizing non-pharmacologic and supportive methods to reduce labor pain is an important part of nursing/midwifery practices. Providing alternatives that allow women to make active decision-making to reduce pain management and anxiety during labor may affect pain, anxiety and hormonal oscillations. Currently, alternative strategies to reduce the use of medication during labor are being considered.

In line with the results of this study, it is thought that the stress ball may be effective in labor, where anxiety and pain are frequently experienced.

After obtaining all official permissions, it is planned to collect the data face-to-face. In the data collection phase, the researcher will first explain the purpose of the study to the women who meet the inclusion criteria and inform them about the study through written consent of the women will be obtained. When the women in the control and experimental groups are admitted to the delivery room, the Introductory Information ; will be collected by the researcher by face-to-face interview method. In addition,;State Anxiety Scale; will be administered during the first admission, VAS before cervical dilatation 0-3 cm, 3-8 cm and 8-10 cm and before placenta emergence, and ;State Anxiety Scale; will be administered when dilatation is 0-3 and 3-8 cm (at the beginning and end of the active phase of labor).;Birth Satisfaction Scale; will be administered in the first 24 hours after delivery before the patient is discharged. Data collection will be done similarly in both groups.

According to randomization, pregnant women in the intervention group will receive ;stress ball therapy; during labor.

ELIGIBILITY:
Inclusion Criteria:

* Being at 38 weeks or more of pregnancy,
* Having a single, healthy fetus in head position,
* Applying during the latent phase of labor (cervical dilatation between 0-3 cm), .To give birth vaginally.

Exclusion Criteria:

* Having become pregnant through assisted reproductive techniques,
* Having a gestational or chronic disease,
* Having an obstacle to giving birth vaginally,
* Suspicion of fetal anomaly,
* Not volunteering to work,
* Women under the age of 18,
* Women who are illiterate in Turkish,
* Decision to perform caesarean section during labor,
* The participant wishes to withdraw from the research,
* Development of fetal distress,
* Using vacuum or forceps during birth, .Women with vision, hearing or mental problems.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Labor pain | Vaginal examination is 0-3 cm in the latent phase, 3-8 cm in the active phase, 8-10 cm in the transitional phase and will be measured with VAS at the end of the second phase and before placenta separation.
  The pregnant woman's pain will be evaluated with VAS.
Anxiety | State anxiety scale will be administered in the latent phase before the stress ball is applied and at 8 cm after the stress ball is applied.
  The state anxiety scale will be filled for anxiety .
Birth satisfaction status | This form will be administered in the first 24 hours after delivery before discharge.
  A minimum of 30 and a maximum of 150 points can be obtained from the scale. The higher the score, the higher the level of satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Karabuk Training and Research Hospital, obstetrics clinic, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No